CLINICAL TRIAL: NCT03847168
Title: Phase I Study of KN026 in HER2 Expressing Breast Cancer, Astric/Gastroesophageal Junction Cancer and Other Locally Advanced/Metastatic Solid Tumors
Brief Title: KN026 in Patients With HER2 Expressing Breast Cancer and Gastric Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN026-US-I-001
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer; Gastric/Gastroesophageal Junction Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KN026 (Experimental): Patient will be intravenously administrated with one dose of KN026. Dosing interval may be adjusted during the study based on emerging data from this trial and/or from other trial.
  Interventions: Drug: KN026

INTERVENTIONS:
Drug: KN026 — Patient will be intravenously administrated with one dose of KN026 every week or every other week.

SUMMARY:
This is an open-label, phase 1 dose-escalation study of KN026 in subjects with HER2 positive advanced breast and Gastric Cancer. The standard "3 + 3" design was used for dose escalation. There are 3 proposed dose levels which are 10, 15, and 20 mg/kg, but dosing interval may be adjusted during the study (such as QW, OR Q2W, OR Q3W) based on emerging data from this trial and/or from phase 1 trial of KN026 in other country. Dose escalation will continue until the maximum tolerated dose (MTD) is reached or if MTD is not found, dose escalation will continue until the MAD of 20 mg / kg is reached.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject >= 18 years
* Histologically/cytologically confirmed, locally advanced unresectable or metastatic breast cancer or gastric cancer.
* ECOG score 0 or 1
* Life expectancy >3 months
* According to the definition of RECIST1.1, the patient has at least one measurable lesion
* Adequate organ function prior to start treatment with KN026
* Able to understand, voluntarily participate and willing to sign the ICF
* Subjects (women of child-bearing potential and males with fertile female partner) must be willing to use viable contraception method.

Exclusion Criteria:

* Accepted any other anti-tumor drug therapies within 4 weeks before fist dose
* Accepted radiotherapy within 4 weeks before enrollment
* An anthracyclines antibiotic treatment was received exceeding 300 mg/m² within 90 days before first KN026 dosing, or other equivalent dose antharcyclines
* Subjects are eligible with clinically controlled and stable neurologic function >= 4 weeks, which is no evidence of CNS disease progression; Subjects with spinal cord compression and cancerous meningitis are not eligible
* Pregnant or nursing females；or intend pregnancy within this study period or within 6 monthes after the end of this study
* History of immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disease, or a history of organ transplantation
* Severe chronic and active infection, need to system antibiosis/antiviral treatment
* Cavity effusion (pleural effusion, ascites, pericardial effusion, etc.) are not well controlled, and need locally treatment or repeated drainage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients experiencing dose limiting toxicities | From screening to up to 28 days

SECONDARY OUTCOMES:
Percentage of participants with adverse events (AEs), serious adverse events (SAEs) and AEs of special interest | From screening to up to 196 days
Maximum observed serum concentration (Cmax) of KN026 | Throughout the duration of the study; up to 84 days
Time of Maximum observed serum concentration (Tmax) of KN026 | Throughout the duration of the study; up to 84 days
Frequency and titer of anti-KN026 antibody | Throughout the duration of the study; up to 2 years
The proportion of patients with an objective response (partial response or complete response) as defined by RECIST 1.1 criteria | Throughout the duration of the study; up to 2 years
Progression free survival according to RECIST 1.1 criteria | Throughout the duration of the study; up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Greenville Health System Center Institute, Greenville, South Carolina, United States